CLINICAL TRIAL: NCT04754958
Title: Evaluation of the Benefit of Virtual Reality to Alleviate Claustrophobia During MRI Clinical Procedure
Brief Title: Virtual Reality to Alleviate Claustrophobia During MRI
Acronym: CLAUSTROVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ecole Polytechnique Fédérale de Lausanne (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Olaf Blanke, Professor Doctor, Ecole Polytechnique Fédérale de Lausanne
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: VRMRI_LNCO2021
Record Dates: First submitted 2021-02-09; First posted 2021-02-15 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Claustrophobia
MeSH Terms: conditions — Claustrophobia | interventions — Immersion

STUDY DESIGN:
Intervention Model Description: Invervention group / no intervention group (standard of care)
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR (Experimental): In addition to standard care during MRI scan, patient receives VR intervention.
  Interventions: Device: Immersion in virtual reality using Nordic Neurolab(™) Visual System
- No VR (No Intervention): Standard of care during MRI scan.

INTERVENTIONS:
Device: Immersion in virtual reality using Nordic Neurolab(™) Visual System — In addition to the standard MRI procedure, the VR intervention group will be looking at stereoscopic computer generated images through a pair of head-coil-mounted googles (Nordic Neurolab ™ Visual System). Two markers (color balls) will be fixed on their knees to capture their movement (camera tracking from the outside of the MRI room). The VR scenario will consist in showing a replication of the actual MRI examination room, as seen from the point of view of the participant lying on the MRI bed, but without the MRI tunnel. Participant can see themselves in the large room (a simplified gender-matched avatar), and an entertaining video can be displayed.
  Arms: VR

SUMMARY:
This study evaluates if our Virtual Reality (VR) simulation inside the MRI efficiently alleviates symptoms of claustrophobia for patients during the MRI examination.

DETAILED DESCRIPTION:
Anxiety of claustrophobic patients during MRI scan leads to movements of patients (which cause imaging artefacts), interruptions or even abortions of imaging scans, eventually requiring to reschedule the examination. Improving these symptoms by creating a VR experiences adapted to the physical constraints of the MRI environment, such as "disappearing the scanner", not only improves the subjective experience of the participant, but has immediate impacts the time spent on the examination, on personnel costs, and resource availability (scanner time).

This study aims at comparing claustrophobic patients in an A|B group design with or without VR intervention. Primary outcomes include subjective reports from patients (Acceptability and Demand) and practitioners (Implementation, Practicality, Adaptation, Integration, Expansion). Secondary outcomes include scanning efficacy based e.g. on the imaging quality, number of times a scan is interrupted by the user and the total duration of a scan. Another non-claustrophobic patients' group will be tested for for obtaining feedback on the general benefit of VR immersion on patients' experience.

ELIGIBILITY:
Inclusion Criteria:

* indicating suffering from claustrophobia
* Be aged between 18 and 40 year-old
* Being able to give consent
* Being able to understand and speak French or English
* Being MRI-compatible

Exclusion Criteria:

* Epilepsy or illnesses affecting the brain, such as HIV, Lyme disease or meningitis
* Psychiatric disorders, such as schizophrenia, autism, obsessive compulsive disorder.
* History of 1 year or more of addiction to drugs such as cannabis, alcohol, cocain, heroine, LSD.
* Taking sleeping pills or anti-anxiety medication before the exam

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Anxiety level | through study completion, an average of one year
  Questionnaire on anxiety during scan (9 items)
Interruption | through study completion, an average of one year
  Record of interruption due to claustrophobia during MRI scan

SECONDARY OUTCOMES:
MRI Image quality | through study completion, an average of one year
  Evaluation of MRI image quality for medical care

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Blanke, Principal Investigator — Ecole Polytechnique Fédéralede Lausanne
Locations (1):
- Hopitaux Universitaires de Geneve (HUG), Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No